CLINICAL TRIAL: NCT02731040
Title: Whole Exome Sequencing to Identify Genetic Predisposition to Atypical Femoral Fractures in Women Using Bisphosphonates for Osteoporosis
Brief Title: Exome Sequencing for Atypical Femoral Fractures
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Steven Mumm, PhD, Associate Professor of Medicine, Washington University School of Medicine
Other Study IDs: 53302
Record Dates: First submitted 2016-03-28; First posted 2016-04-07 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Atypical Femoral Fractures; Osteoporosis; Bisphosphonate Therapy
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates; Alendronate; Zoledronic Acid; Risedronic Acid; Etidronic Acid; Ibandronic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Controls: Women who are/have been on bisphosphonate therapy for osteoporosis who have not suffered an atypical femoral fracture
  Interventions: Drug: Bisphosphonate
- Fracture Group: Women who are/have been on bisphosphonate therapy for osteoporosis who have suffered an atypical femoral fracture
  Interventions: Drug: Bisphosphonate

INTERVENTIONS:
Drug: Bisphosphonate
  Other Names: Aledronate (Fosamax); Zoledronate (Zometa and Reclast); Risendronate (Actonel and Atelvia); Etidronate (Didronel); Ibandronate (Boniva)

SUMMARY:
The purpose of this study is to determine whether women who have atypical subtrochanteric and diaphyseal femoral fractures after treatment with bisphosphonates for osteoporosis, have a genetic predisposition to these unusual fractures.

DETAILED DESCRIPTION:
In 2010, a Task Force convened by the American Society for Bone and Mineral Research (ASBMR) investigated an apparent association of atypical subtrochanteric and diaphyseal femoral fractures (AFFs) with long-term bisphosphonate (BP) treatment given for the important and common disorder osteoporosis (OP).(1,2) Because the investigators had reported(2) in 2009 that the prodromal lesion for AFFs in OP resembles the femoral pseudofractures encountered in the rare adult form of hypophosphatasia (HPP),(3-5) they recommended sequencing the tissue non-specific alkaline phosphatase (TNSALP) gene of OP AFF patients to determine if mutations or polymorphisms in TNSALP genetically predispose to OP AFFs.(2)

In 2012, the investigators reported a 55-year-old woman treated for four years with BPs for presumed OP who then suffered simultaneous atraumatic bilateral AFFs.(4) Upon sequencing her TNSALP, a heterozygous mutation changing an arginine (Arg) to a histidine (His) (c.212 G>A, p.Arg71His) was discovered that the investigators had documented in the investigators' large cohort of HPP patients. She had been undiagnosed with HPP although her pre-BP serum ALP was persistently low (26 U/L, Nl 32 - 116 U/L). The investigators then recruited and sequenced TNSALP for 24 new OP AFF patients given BPs, and identified a second OP AFF patient carrying a TNSALP defect.(3) These two OP AFF patients with TNSALP defects support the investigators' hypothesis (below) that high-impact rare genetic variants in TNSALP, and perhaps other genes, can predispose to OP AFFs.(4) Furthermore, the investigators reported in 2009(2) that the prodromal lesions of OP AFFs can resemble the femoral pseudofractures seen in another, but more prevalent, heritable metabolic bone disease, X-linked hypophosphatemia (XLH). This is the most common genetic cause of osteomalacia,(6) and is inherited as an X-linked dominant trait caused by deactivating mutations in the PHEX gene.

Osteoporosis (OP) is a complex disorder likely involving the effects of multiple low-impact, common changes in the human genome that alter bone remodeling and/or mineralization.(7-9) The investigators propose that high-impact, rare, genetic variants predispose some OP patients to AFFs. Treatment with BPs could engender OP AFFs. The investigators' hypothesis: High-impact rare variants (i.e., mutations) that occur in genes/proteins that regulate pyrophosphate/phosphate homeostasis or BP metabolism predispose to OP AFFs and are unmasked in OP patients given BPs. Identification of these variants will guide OP therapies, perhaps on an individual basis (i.e., "personalized medicine"),(9) and reduce the incidence of OP AFFs.

The investigators will identify high-impact rare genetic variants using whole exome sequencing in two patient groups: 1) women using BPs for OP and have had one or more AFF, 2) women using BPs for OP but have not had an AFF. The investigators will focus on genes/proteins that: i) regulate pyrophosphate/phosphate effects, ii) others that regulate BP metabolism, and iii) have been associated with OP. The investigators will use gene burden analysis to determine whether there is an excess of novel or rare genetic variants for the group with AFFs.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Previous and/or current use of bisphosphonate therapy for the management of osteoporosis

For inclusion in the fracture group must have:

-sustained one or more atypical subtrochanteric or diaphyseal femoral shaft fracture(s) as defined by the the 2010 ASBMR task force.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who are or have been taking bisphosphonates for osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Whole Exome Sequencing to identify mutations in genes that regulate pyrophosphate metabolism. | Within the first year of study
  Whole Exome Sequencing will be used to identify changes in DNA sequences of genes which regulate pyrophosphate metabolism. These changes could alter the amino acid sequence, and may include termination of translation, or affect mRNA splicing.
Whole Exome Sequencing to identify mutations in genes that regulate phosphate metabolism. | Within the first year of study
  Whole Exome Sequencing will be used to identify changes in DNA sequences of genes which regulate phosphate metabolism. These changes could alter the amino acid sequence, and may include termination of translation, or affect mRNA splicing.
Whole Exome Sequencing to identify mutations in genes that regulate bisphosphonate metabolism. | Within the first year of study
  Whole Exome Sequencing will be used to identify changes in DNA sequences of genes which regulate bisphosphonate metabolism. These changes could alter the amino acid sequence, and may include termination of translation, or affect mRNA splicing.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Mumm, PhD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Shane E, Burr D, Ebeling PR, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster D, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Koval K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Sen HT, van der Meulen MC, Weinstein RS, Whyte M; American Society for Bone and Mineral Research. Atypical subtrochanteric and diaphyseal femoral fractures: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2010 Nov;25(11):2267-94. doi: 10.1002/jbmr.253. PMID 20842676
- [Background] Shane E, Burr D, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster DW, Ebeling PR, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Howe TS, van der Meulen MC, Weinstein RS, Whyte MP. Atypical subtrochanteric and diaphyseal femoral fractures: second report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2014 Jan;29(1):1-23. doi: 10.1002/jbmr.1998. Epub 2013 Oct 1. PMID 23712442
- [Background] 2013 Annual Meeting of the American Society for Bone and Mineral Research, October 4-7, 2013, Baltimore, MD. J Bone Miner Res. 2013 Feb;28 Suppl 1:S1. doi: 10.1002/jbmr.2201. No abstract available. PMID 24585702
- [Background] Sutton RA, Mumm S, Coburn SP, Ericson KL, Whyte MP. "Atypical femoral fractures" during bisphosphonate exposure in adult hypophosphatasia. J Bone Miner Res. 2012 May;27(5):987-94. doi: 10.1002/jbmr.1565. PMID 22322541
- [Background] Whyte MP. Hypophosphatasia. In Pediatric Bone: Biology & Diseases, 3rd ed. Glorieux FH, Jueppner H, Pettifor J, eds. San Diego, CA: Elsevier, 2012;771-794.
- [Background] Reid IR, Hardy DC, Murphy WA, Teitelbaum SL, Bergfeld MA, Whyte MP. X-linked hypophosphatemia: a clinical, biochemical, and histopathologic assessment of morbidity in adults. Medicine (Baltimore). 1989 Nov;68(6):336-52. PMID 2811660
- [Background] Duncan, E.L., Brown, M.A. Genome-wide association studies (2013) Genetics of Bone Biology and Skeletal Disease, pp. 93-100
- [Background] Nguyen, T.V., Eisman, J.A. Pharmacogenetics and pharmacogenomics of osteoporosis: personalized medicine outlook (2013) Genetics of Bone Biology and Skeletal Disease, pp. 151-167
- [Background] Rivadeneira, F., Uitterlinden, A.G. Osteoporosis Genes Identified by Genome-wide Association Studies (2013) Genetics of Bone Biology and Skeletal Disease, pp. 243-256.